CLINICAL TRIAL: NCT00611221
Title: Massage Therapy and Labour Outcomes; A Randomized Controlled Trial
Brief Title: Massage Therapy Study: Massage Therapy and Labour Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Massage Therapy Foundation (Other); Holistic Health Research (Unknown)
Responsible Party: Patricia Janssen, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H07-00528; CW07-0090
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Pain During Labour
Keywords: massage; labour
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Massage therapy by a regulated massage therapist
  Interventions: Procedure: Massage
- 2 (Active Comparator): Massage by anyone else, eg. husband, nurse, doula
  Interventions: Procedure: Massage

INTERVENTIONS:
Procedure: Massage — Massage therapy by an RMT during labour
  Arms: 1
Procedure: Massage — Massage by anyone else, eg. husband, nurse, doula
  Arms: 2

SUMMARY:
OBJECTIVE: To measure the benefits of massage, administered by a registered massage therapist, to pain management for women in active labour.

DESIGN: A randomized controlled trial.

SETTING: BC Women's Hospital, a tertiary level maternity teaching hospital in Vancouver, British Columbia, Canada.

PARTICIPANTS: Healthy first time mothers experiencing an uncomplicated pregnancy who present to the hospital in labour. Seventy women will be enrolled in each trial arm.

MAIN OUTCOME MEASURES: The primary outcome is time to use of epidural analgesia measured as cervical dilatation at the time of epidural insertion. Secondary outcomes include use of epidural and narcotic analgesia, and measures of intensity and characteristics of pain.

DATA ANALYSIS: Study outcomes will be compared among women randomized to receive a maximum of five hours of massage during labour administered by a registered massage therapist versus usual care. Analysis will be by intention to treat. Prognostics factors not balanced between trial arms (massage and usual care) will be controlled for in a multivariate analysis.

DETAILED DESCRIPTION:
Goal and Objectives:

The overall purpose of this project is to evaluate the effectiveness of massage therapy provided by registered massage therapists in managing pain among women in active labour.

Specific Aims:

Our specific aim is to randomly assign women admitted to hospital in active labour to receive a maximum of five hours massage by a regulated massage therapist or usual care in order to study the effect of massage therapy on pain relief, labour management and patient outcomes.

Research Questions:

We will compare among healthy, nulliparous women experiencing health pregnancies with access to massage therapy after admission to hospital in active labour vs. women receiving usual care:

* the severity and quality of pain from contractions
* among women carrying a fetus in the occiput posterior position, the severity of back pain
* length of first and second stage of labour
* need for use of entonox, sterile water injections, intravenous or intramuscular narcotics, and epidural analgesia
* stage of labour (cervical dilatation) among those women who receive epidural analgesia
* position of occiput at the onset of second stage
* mode of delivery: spontaneous vaginal, assisted (vacuum/forceps), and caesarean section
* time to first breastfeeding after delivery

Hypotheses:

We hypothesize that healthy women who receive massage therapy during active labour will:

* at a given cervical dilatation, experience less severe pain with contractions
* if carrying a fetus in the occiput posterior position, at a given cervical dilatation, will report less severe back pain
* experience a shorter first and second stage of labour
* be more likely to request entenox
* be more likely to request sterile water injections
* be more likely to request intravenous or intramuscular narcotics
* be less likely to request epidural analgesia
* if requesting epidural analgesia, to request it at a later stage (greater cervical dilatation) in labour
* The fetal occiput will be more likely to be anterior vs. posterior at the onset of second stage of labour
* be less likely to deliver by caesarean section
* undertake their first breastfeeding more quickly after delivery

Design:

We propose a randomized two-arm unblinded controlled trial. The treatment condition is massage therapy during the active phase of labour by a registered massage therapist. The control condition is usual care. The primary outcome is cervical dilatation at request for epidural analgesia.

Study sample:

Our study sample will be drawn from healthy nulliparous women experiencing healthy pregnancies presenting for intrapartum care at BC Women's Hospital.

Study Setting:

The study will take place at BC Women's Hospital in Vancouver, British Columbia, Canada. BC Women's is an academic teaching hospital. It provides primary care to women who are residents of the City of Vancouver, regional referral care to residents of the Lower Mainland or southwest corner of the province, and tertiary referral care for the entire province. Approximately 7500 take place at this hospital annually; about 7000 are to women who reside in Vancouver. All women for whom delivery is not imminent are triaged in a large assessment room adjacent to the delivery suite prior to being admitted for intrapartum care. Women in labour have one-to-one care in a private labour room. They may have whomever else they want in the room to support them.

Recruitment:

Women will be approached for participation in the study by a registered, experienced obstetrical nurse on admission to the assessment area of the hospital. At present, this service is provided by the Maternal/fetal Medicine Division of the Department of Obstetrics and Gynecology, for a fee.

Randomization:

Randomization will take place immediately after obtaining written consent. A statistical software package (SPSS - Statistical Program for the Social Sciences) will be utilized to randomly assign sequential numbers to one of the two treatment arms. Cards will be numbered sequentially and labelled with the treatment allocation. These cards will be placed in opaque envelopes in a box which will be kept in a locked cupboard to which the recruitment nurse holds the key. Envelopes will be opened in sequential order for each study participant after written informed consent has been obtained. A log book will be maintained by the recruitment nurse detailing the patients approached, their decision to participate or not, randomization number, and allocation.

Protocol:

Immediately after randomization, the recruitment nurse will contact the massage therapist on call by means of a cell phone. Massage therapists named in this application have agreed to be on call for the study for periods in total that cover 7 days per week. The massage therapist will leave immediately to come and provide massage therapy. The massage therapist will receive a brief report from the women's labour and delivery nurse as to what nature of the woman's labour to that point. She will then explain to the women what she would suggest for specific massage techniques and will begin as soon as the woman is ready. It should be noted that women may continue to use other non-invasive pain management modalities as they wish. This is a pragmatic trial in that massage therapy is seen as one additional choice that women will have access to in addition to the repertoire of choices that are routinely available.

Study Outcomes:

Our primary outcome is timing of epidural analgesia with respect to cervical dilatation. This outcome is chosen because 67% of nulliparous women at this institution have epidural analgesia and because of the association of epidural use with intrapartum interventions. In the current study we would like to be able to detect a mean decrease in cervical dilation at the time of request for epidural as small as 1 cm. In order to find a decrease of 1 cm in cervical dilation, which is a clinically important difference, we would need 42 study subjects per group with 80% power and a type I error set at p =.05, one sided. Since we learned from our previous study that 61% of women meeting study inclusion criteria receive an epidural prior to 10 cm dilatation, we know that we will have to recruit 70 women per study arm to have 42 people in each arm who receive an epidural.

ELIGIBILITY:
Inclusion Criteria:

* Healthy primiparous women
* Nulliparous
* Singleton gestation
* Cephalic presentation
* Term gestation (37-41 completed weeks of pregnancy)
* Maternal age between 18 and 35 years of age
* In spontaneous labour, defined for our purposes as painful contractions which have resulted in cervical change, i.e. cervix is 1 cm dilated or more with effacement at 25% (0.5 cm) or more on admission to the labour unit
* Able to speak and read English or speak a language for which there is a nursing interpreter available

Exclusion Criteria

* Pre-existing medical conditions including but not limited to: insulin dependent diabetes, renal, cardiac, or thyroid conditions, hypertension, epilepsy, psychosis, use of illicit street drugs
* Conditions arising during pregnancy which require non-routine surveillance and/or intervention including but not limited to gestational diabetes, gestational hypertension, 2nd or 3rd trimester hemorrhage, intrauterine growth restriction, presence of a fetal congenital anomaly, history of preterm prelabour rupture of membranes
* Statement by women on admission that she has been in labour for more than 24 hours
* Cervical dilatation 10 cm (full dilatation) on admission to the labour ward

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is time to use of epidural analgesia measured as cervical dilatation at the time of epidural insertion. | During labour

SECONDARY OUTCOMES:
Secondary outcomes include use of epidural and narcotic analgesia and measures of intensity and characteristics of pain. | During labour

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Janssen, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada